CLINICAL TRIAL: NCT01262742
Title: Carbetocin at Elective Cesarean Delivery: A Dose Finding Study
Brief Title: Carbetocin at Elective Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-02
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2011-09

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; Cesarean delivery; carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Carbetocin 80mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 90mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 100mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 110mcg (Active Comparator)
  Interventions: Drug: Carbetocin
- Carbetocin 120mcg (Active Comparator)
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — 80mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 80mcg
Drug: Carbetocin — 90mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 90mcg
Drug: Carbetocin — 100mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 100mcg
Drug: Carbetocin — 110mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 110mcg
Drug: Carbetocin — 120mcg carbetocin, IV, over 1 minute following delivery of the fetal head.
  Other Names: Duratocin
  Arms: Carbetocin 120mcg

SUMMARY:
Post-partum hemorrhage (PPH) is a major cause of maternal death worldwide. Oxytocin is the most commonly uterotonic drug used to prevent and treat PPH in North America, however, there are some limitations to its use. Oxytocin has a very short duration of action, which requires a continuous infusion to achieve sustained uterotonic activity. The Society of Obstetricians and Gynecologists of Canada (SOGC) has recently recommended a single 100mcg dose of carbetocin at elective Cesarean delivery to promote uterine contraction and prevent post partum hemorrhage (PPH), in lieu of the more traditional oxytocin regimens. Carbetocin lasts 4 to 7 times longer than oxytocin, with a similar side effect profile and apparent greater efficacy rate. However, a dose response to determine the minimum effective dose of carbetocin has not yet been published.

We hypothesize that a dose-response study will establish the minimum dose of carbetocin required to produce appropriate contractility in 95% of the women (ED95) undergoing elective cesarean delivery.

DETAILED DESCRIPTION:
The Society of Obstetricians and Gynecologists of Canada (SOGC)recently recommended a 100mcg intravenous bolus dose of carbetocin following Cesarean delivery. However, a dose response study to determine the minimum effective dose of carbetocin has not yet been published.

Studies thus far show that carbetocin may be just as effective as oxytocin in promoting uterine contraction, with a similar side effects profile. In addition, patients receiving carbetocin may experience less blood loss, and require less additional uterotonics when compared with oxytocin.

The results of this study will define the minimum required dose of carbetocin for uterine contraction, thus minimizing unnecessary side effects, improving quality and safety of patient care. It may also contribute in establishing carbetocin as a substitute to oxytocin for elective cesarean section at our institution as well as others.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for elective cesarean delivery under spinal anesthesia;
* All patients who gave written informed consent to participate in this study.

Exclusion Criteria:

* All patients who refuse to give written informed consent.
* All patients who claim allergy or hypersensitivity to carbetocin or oxytocin.
* All patients with conditions that predispose to uterine atony and postpartum hemorrhage such as placenta previa, multiple gestation, preeclampsia, eclampsia, macrosomia, polyhydramnios, uterine fibroids, previous history of uterine atony and postpartum bleeding, or bleeding diathesis.
* All patients with hepatic, renal, and vascular disease,
* All patients requiring general anesthesia prior to the administration of the study drug.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Uterine tone. | 2 minutes
  The obstetrician will assess uterine tone by palpation. Uterine tone will be rated as satisfactory (firm) or unsatisfactory (boggy).

SECONDARY OUTCOMES:
Uterine tone | 2 hours
  Uterine tone will be assessed by palpation 2 hours post-delivery by the nurse/obstetrician in the recovery room.
Blood loss | 48 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 48 hours after the cesarean section.
Side effects | 2 hours
  Any of the following will be noted up to 2 hours post delivery: systolic blood pressure < 80% of pre-delivery values, tachycardia > 30% pre-delivery levels, bradycardia < 30% pre-delivery levels, other dysrhythmias, nausea, vomiting, chest pain, shortness of breath, headache, flushing, others

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cordovani D, Balki M, Farine D, Seaward G, Carvalho JC. Carbetocin at elective Cesarean delivery: a randomized controlled trial to determine the effective dose. Can J Anaesth. 2012 Aug;59(8):751-7. doi: 10.1007/s12630-012-9728-2. Epub 2012 Jun 21. PMID 22717890